CLINICAL TRIAL: NCT02629939
Title: Basic Knowledge of CPR Among Close Relatives of Heart Patients-check Status Quo and Attemp to Establish a Potential Plan to Implement This Knowledge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Yan Press, family medicine , Ben Gurion University of the Negev, Meir Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0136-15-COM1
Record Dates: First submitted 2015-12-02; First posted 2015-12-15 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Cardiopulmonary Resuscitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- questionnaires (No Intervention): Questionnaires will be distributed to families of heart patients to test the theoretical knowledge to perform CPR The questionnaires were distributed to internal, cardiology clinics and clinic T by a doctor, Paramedic or medical student. The family will be asked to fill out the questionnaire independently.
  The questionnaires will be distributed in Hebrew, Arabic, Russian and English The research questionnaire will include questions about able to perform basic CPR
- to participate in a short course for learning CPR (Experimental): : The investigators will offer patients and their relatives to participate in a short course for learning CPR.
  Relatives will receive a "prescription" Containing a proposal for participation in the course
  Prescription will be awarded in four places:
  -.Family physicians as a suggestion during a routine visit / presentation of cardiac problem
  * Heart Rehabilitation Institute - "cardionegev"
  * Doctors internal medicine department as part of a patient's discharge letter with heart disease
  * Doctors in cardiology clinic The prescription will be accompanied by several minutes of explanation about the program and its importance The investigators consider the level of responsiveness and participation, find out which arm yielded the highest number of participants (actual turnout of the total prescriptions distributed) And how to expand their activities
  Interventions: Behavioral: course for learning CPR

INTERVENTIONS:
Behavioral: course for learning CPR
  Arms: to participate in a short course for learning CPR

SUMMARY:
Cardiac arrest is a public health problem and is the leading cause of death in many parts of the world.

Cardiac arrest can occur inside the hospital and outside it. In the United States and Canada occur in approximately 350,000 cases of cardiac arrest a year , who receive CPR , Half of them outside the hospital.

Treatment of cardiac arrest is performing Cardio Pulmonary Resuscitation (CPR) and early defibrillation.

Performing compressions is the essential part of performing CPR until the arrival of defibrillation.

Efforts are being made to simplify the implementation of basic CPR and make it accessible to everyone. Method "hands only CPR" offers CPR with compressions only without ventilations, Studies have shown a similar survival rate between" hands only CPR" method and CPR with ventilations.

Patient's chances of survival are higher if a bystander begins performing CPR until trained medical staff arrives.

Chances of survival decreases by 7-10% every passing minute past moment of collapse if not performed CPR.

MDA survey carried out in 1984-5 reported at the start of CPR by a bystander at 8% Another survey in 2000 reported 14%, In a recent study in Jerusalem found a rate of only 15% of performing compressions by bystanders- A very low rate compared to 33% reported in the United States 41.3% in Japan and 44.9% in Denmark.

The average time of arrival of the medical team in Israel is 10.3 minutes, so it is very important to begin performing CPR by those present before the arrival of medical staff.

Most cases of cardiac arrest were the result of a previous cardiac disease, Therefore patients with cardiac disease are at higher risk of cardiac arrest and cardiac death.

Place cardiac arrest is 72% percent of the time at home, and the likely presence of family members.

The general population should know basic resuscitation to save a life, knowledge is needed especially among families of heart patients who are way more likely that such an event will occur in their presence.

Therefore, one can relate to families of heart patients dedicated to increasing population as a basic knowledge of CPR.

There is no other organized plan to study family members of patients with heart disease basic knowledge of CPR Despite the importance of it Attempts have been published in previous studies from around the world to create a focus group study of CPR among close relatives of heart patients. An attempt was made to incorporate as part of the proposed cardiac rehabilitation patients after MI Through self-study kit given at discharge from the hospital and more Difficult to evaluate the success of these efforts over the long term, but short-term study of short workshops yielded sufficient knowledge about basic CPR This study should serve as a catalyst as a first step towards building a suitable program nationwide and hopefully save many lives

DETAILED DESCRIPTION:
Cardiac arrest is a public health problem and is the leading cause of death in many parts of the world.

Cardiac arrest can occur inside the hospital and outside it. In the United States and Canada occur in approximately 350,000 cases of cardiac arrest a year , who receive CPR , Half of them outside the hospital.

Treatment of cardiac arrest is performing Cardio Pulmonary Resuscitation (CPR) and early defibrillation.

Performing compressions is the essential part of performing CPR until the arrival of defibrillation.

Efforts are being made to simplify the implementation of basic CPR and make it accessible to everyone. Method "hands only CPR" offers CPR with compressions only without ventilations, Studies have shown a similar survival rate between" hands only CPR" method and CPR with ventilations.

Patient's chances of survival are higher if a bystander begins performing CPR until trained medical staff arrives.

Chances of survival decreases by 7-10% every passing minute past moment of collapse if not performed CPR.

MDA survey carried out in 1984-5 reported at the start of CPR by a bystander at 8% Another survey in 2000 reported 14%, In a recent study in Jerusalem found a rate of only 15% of performing compressions by bystanders- A very low rate compared to 33% reported in the United States 41.3% in Japan and 44.9% in Denmark.

The average time of arrival of the medical team in Israel is 10.3 minutes, so it is very important to begin performing CPR by those present before the arrival of medical staff.

Most cases of cardiac arrest were the result of a previous cardiac disease, Therefore patients with cardiac disease are at higher risk of cardiac arrest and cardiac death.

Place cardiac arrest is 72% percent of the time at home, and the likely presence of family members.

The general population should know basic resuscitation to save a life, knowledge is needed especially among families of heart patients who are way more likely that such an event will occur in their presence.

Therefore, one can relate to families of heart patients dedicated to increasing population as a basic knowledge of CPR.

There is no other organized plan to study family members of patients with heart disease basic knowledge of CPR Despite the importance of it Attempts have been published in previous studies from around the world to create a focus group study of CPR among close relatives of heart patients. An attempt was made to incorporate as part of the proposed cardiac rehabilitation patients after MI Through self-study kit given at discharge from the hospital and more Difficult to evaluate the success of these efforts over the long term, but short-term study of short workshops yielded sufficient knowledge about basic CPR This study should serve as a catalyst as a first step towards building a suitable program nationwide and hopefully save many lives

ELIGIBILITY:
Inclusion Criteria:

* over 18
* Insured by Clalit Health Services only
* First-degree relatives or those living with the patient in the same house
* The course will be for Hebrew -speaking only

Exclusion Criteria:

* Under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
CPR knowledge from self-administrated questionnaire | up to one month before CPR course
CPR knowledge from self-administrated questionnaire | 3 months after CPR course

CONTACTS AND LOCATIONS:
Locations (1):
- Yan Press, Beersheba, Israel